CLINICAL TRIAL: NCT05975814
Title: Effect of the Shape of the Healing Abutment on Soft Tissue Healing. A Randomized Clinical Study Involving an Enhanced Digital Superposition Methodology
Brief Title: The Effect of Concave Healing Abutment on Soft Tissue Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MIS Implant Technologies, Ltd (Industry)
Collaborators: Charite University, Berlin, Germany (Other); Sachsen Praxen Zahnarztpraxis (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIS-CONCAVE
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Dental Implant Therapy
Keywords: dental implants; concave abutments; intra-oral scans; CBCT; soft tissue thickness; randomized clinical study
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: clinical study
Masking Description: each implant receives either a straight or a concave abutment. The patient is not aware of the type of abutment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- concave abutment vs. straight abutment (Experimental): After implant is placed a randomization will determine if the implant receives a straight or a concave abutment. If a patient requires 2 implants, one of them will be straight and the other will be concave. A patient can therefore have both abutments.
  Interventions: Device: dental implant

INTERVENTIONS:
Device: dental implant — dental implants are placed as usual and require a healing abutment. Abutments can be straight or concave, both are equally available on the market.

SUMMARY:
The aim of this study is to document the relevance of the concave abutment to form more gingiva when compared to the straight abutment.

DETAILED DESCRIPTION:
Standard clinical and radiographic examination will assess the need for implant therapy, the number of implants and the rehabilitation type. The pre-operative skeletal data will be observed with a 3D cone-beam computed tomographic examination (Cranex 3D, Soredex, Tuusula, Finland). On implantation day just before surgery, an initial intra-oral scan (TRIOS3, 3Shape, Copenhagen, Denmark) will be taken (IOS#0) to provide the baseline of the soft tissue outline. The surgical procedure will involve a crestal incision with 2 lateral discharge incisions; a full flap will be raised and the periosteum will be carefully separated from the cortical bone. The implant osteotomy will be prepared by executing the drilling sequence recommended by the manufacturer according to bone density; the final single-use drill that comes with each implant will be implemented on top of the drills when relevant. SEVEN (MIS) Ø 4.2 mm implants with an internal hex connection of appropriate length will be placed according to a 1-stage surgical protocol. They will receive a Ø 4.8 x 6 mm wide abutment, either straight or concave, according to the randomization. To anticipate early bone loss the implants will be seated slightly in a subcrestal position.

For single crown rehabilitations, a coin randomization will be performed to determine the abutment type, straight or concave; for plural restorations, randomization will start from the most distal implant. Height of all healing abutments will be 6 mm because this item provides the largest available mismatch concavity, 0.6 mm, compared to the straight abutment. After implant and abutment placement, the flap and periosteum will be reclined and sutured with single discontinued sutures around the abutments without tension. The patients will receive antibiotics (875/125 mg of Amoxicillin/Clavulanic acid, 3/d for 7 days; in case of penicillin allergy, 300 mg of Clindamycin every 6 h for 7 days) and analgesic anti-inflammatory treatment (600 mg Ibuprofen 3/d); rinsing with Chlorhexidine (0.12%) (Dentaid® PerioAid 0.12%) will be prescribed 2/d for 2 weeks. Sutures will be removed after 10 days (Cacaci et al., 2021). After a transmucosal soft tissue healing period of 6-8 weeks, the healed sites will be scanned (IOS#1).

ELIGIBILITY:
Inclusion Criteria:

a) patients older than 18 years in need of implant therapy in the posterior area of the mandible and maxilla, b) good general/systemic health (ASA type I, II), c) patients who committed to attend all visits of the study, d) placement of a Ø 4.2 mm implant without requiring bone augmentation, e) adequate oral hygiene with FMPS (full mouth plaque score) < 15% before surgery, f) absence of uncontrolled periodontal disease, g) agreeing to sign an informed consent.

Exclusion Criteria:

a) patients with a contributing medical history in which any surgery, disease, condition, or medication susceptible to compromise the healing of soft and hard tissues (e.g. non-controlled diabetes), b) liver function disorder, c) immune system disease, d) immunosuppressant drugs, e) toxic habits other than smoking that might compromise or affect healing, f) patients who have undergone chemotherapy or radiation treatment during the previous 5 years comprising the head and neck area, g) corticosteroids therapy or any other medication that could influence postoperative healing and/or osseointegration, h) bisphosphonate or Denosumab therapy (Prolia®), i) sites that underwent or require a horizontal or vertical bone regeneration procedure, j) inability or unwillingness to attend follow-up visits, k) patients unwilling to sign an informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Thickness of the peri-implant gingiva at the level of the largest mismatch between the straight and the concave abutment | end of healing, 6-8 weeks after implant surgery
  The thickness of the gingiva will be measured on the superposition set including the STL of the abutments on the vestibular and lingual/palatal sides

SECONDARY OUTCOMES:
Height of the peri-implant gingiva at the level of the largest mismatch between the straight and the concave abutment | end of healing, 6-8 weeks after implant surgery
  The height of the gingiva will be measured on the superposition set including the STL of the abutments on the vestibular and lingual/palatal sides

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Sperber, Dr, Principal Investigator — Sachen Praxen
Locations (1):
- Mis Implants Technologies Ltd., Misgav Regional Council, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lilet R, Desiron M, Finelle G, Lecloux G, Seidel L, Lambert F. Immediate implant placement combining socket seal abutment and peri-implant socket filling: A prospective case series. Clin Oral Implants Res. 2022 Jan;33(1):33-44. doi: 10.1111/clr.13852. Epub 2021 Oct 22. PMID 34551159